CLINICAL TRIAL: NCT03015506
Title: Measuring the Glycemic Index of Pulse Based Breads
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glycemic Index Laboratories, Inc (Industry)
Collaborators: Agriculture and Agri-Food Canada (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 01E91-16-62508
Record Dates: First submitted 2017-01-06; First posted 2017-01-10 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-01

CONDITIONS: Carbohydrate Intolerance
MeSH Terms: conditions — Glucose-Galactose Malabsorption | interventions — Bread

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- White Bread (Active Comparator): Portion of bread containing 50g available carbohydrate (defined as total carbohydrate minus dietary fiber).
  Interventions: Other: Bread
- Pea Bread (Experimental): Portion of bread containing 50g available carbohydrate (defined as total carbohydrate minus dietary fiber) containing 18% (by weight) pea flour.
  Interventions: Other: Bread
- Green Lentil Bread (Experimental): Portion of bread containing 50g available carbohydrate (defined as total carbohydrate minus dietary fiber) containing 18% (by weight) green lentil flour.
  Interventions: Other: Bread
- Red Lentil Bread (Experimental): Portion of bread containing 50g available carbohydrate (defined as total carbohydrate minus dietary fiber) containing 18% (by weight) red lentil flour.
  Interventions: Other: Bread
- Chickpea Bread (Experimental): Portion of bread containing 50g available carbohydrate (defined as total carbohydrate minus dietary fiber) containing 18% (by weight) chickpea flour.
  Interventions: Other: Bread

INTERVENTIONS:
Other: Bread

SUMMARY:
The objective of this study is to determine the glycemic index of 4 pulse-based breads in at least 10 normal healthy human volunteers. Participants will be studied in the morning on 6 separate days after overnight fasts. On the first and last days they will consume a test meal consisting of about 2 slices of white bread (50g carbohydrate) and on the other 4 days they will consume 2-3 slices (50g carbohydrate) from 4 different test breads containing starch obtained from pulses (beans and/or lentils). Blood glucose will be measured at intervals over 2 hours. Glycemic index is calculated as 0.71 times F/WB where F is the incremental area under the curve of blood glucose (AUC) after each test bread and WB is the mean AUC after white bread.

ELIGIBILITY:
Inclusion Criteria:

* participants in good health

Exclusion Criteria:

* known history of HIV
* known history of diabetes
* history of hepatitis within the last 3 months
* heart condition requiring hospitalization within 3 months
* use of medications or presence of any condition which in the opinion of the study physician, would increase the risk of harm to the subject or to others, or affect the results of the study.
* participants who cannot or will not comply with experimental procedures or the safety guidelines of Glycemic Index Laboratories, Inc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Glycemic Index | 120 minutes
  Glycemic index is 0.71 times F/WB where F is the incremental area under the blood glucose response curve ignoring area below fasting (AUC) elicited by a pulse bread, and WB is the mean AUC elicited by White Bread. AUC is calculated using the trapezoid rule from 2 measures of fasting blood glucose taken 5 minutes apart (the average of these measures is taken to be fasting blood glucose) and measures of blood glucose at 15, 30, 45, 60, 90 and 120 minutes after starting to eat. The mean of the values for each pulse bread in each subject is the glycemic index.

SECONDARY OUTCOMES:
Incremental area under the blood glucose response curve | 120 minutes
  Incremental area under the blood glucose response curve ignoring area below fasting (AUC) is calculated using the trapezoid rule from 2 measures of fasting blood glucose taken about 5 minutes apart (the average of these measures is taken to be fasting blood glucose) and measures of blood glucose at 15, 30, 45, 60, 90 and 120 minutes after starting to eat.
Peak blood glucose concentration (Cmax) | 120 minutes
  Cmax is the maximum of the blood glucose concentrations measured at 15, 30, 45, 60, 90 and 120 minutes after consumption of a test meal.
Peak rise of blood glucose | 120 minutes
  The maximum of the blood glucose concentrations measured at 15, 30, 45, 60, 90 and 120 minutes after consumption of a test meal minus the fasting blood glucose concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, MD, PhD, Principal Investigator — Glycemic Index Laboratories, Inc

IPD SHARING:
Plan to Share IPD: No